CLINICAL TRIAL: NCT04887610
Title: Factors That Influence Blood Vessel Regulation During Exercise in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Philip Millar, Associate Professor, University of Guelph
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20-11-008
Record Dates: First submitted 2021-04-01; First posted 2021-05-14 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Ischemic Preconditioning; Dietary Exposure
MeSH Terms: interventions — Ischemic Preconditioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ischemic preconditioning control (Sham Comparator)
  Interventions: Procedure: Ischemic preconditioning control
- Ischemic preconditioning (Active Comparator)
  Interventions: Procedure: Ischemic preconditioning
- High fat meal (Active Comparator)
  Interventions: Dietary Supplement: Low fat meal
- Low fat meal (Placebo Comparator)
  Interventions: Dietary Supplement: High fat meal

INTERVENTIONS:
Procedure: Ischemic preconditioning — Four 5-minute cycles of 200 mmHg cuff inflation of the brachial artery, each separated by 5-minutes deflated recovery (i.e. 40 minutes total time)
  Arms: Ischemic preconditioning
Procedure: Ischemic preconditioning control — Four 5-minute cycles of 20 mmHg cuff inflation of the brachial artery, each separated by 5-minutes deflated recovery (i.e. 40 minutes total time)
  Arms: Ischemic preconditioning control
Dietary Supplement: Low fat meal — Meal containing 1006 calories, 1 g fat, 0.2 g saturated fat, 0 g trans fat, 20 mg cholesterol, 191 g carbohydrates, 60 g protein, 1560 mg sodium
  Arms: High fat meal
Dietary Supplement: High fat meal — Meal containing 1030 calories, 62 g fat, 23 g saturated fat, 0.5 g trans fat, 445 mg cholesterol, 76 g carbohydrates, 41 g protein, 2080 mg sodium.
  Arms: Low fat meal

SUMMARY:
This study will examine two separate interventions: 1) the effects of ischemic preconditioning or 2) a high fat meal on the capacity of the brachial artery to overcome sympathetic activation and dilate during exercise (also known as functional sympatholysis). Participants will be asked to complete rhythmic handgrip exercise with and without the application of -20 mmHg lower body negative pressure to increase sympathetic activation. Doppler ultrasound will be used to continuously measure brachial artery blood flow. Participants will complete the handgrip exercise and lower body negative pressure before and after the applications of each interventions. Participants may elect to only complete one intervention rather than complete both protocols. Intervention one is active or control ischemic preconditioning. Intervention two is high or low fat meals.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Healthy

Exclusion Criteria:

* History of smoking (tobacco or cannabis), defined as any smoking within the past 3 months
* Diagnosed cardiovascular or metabolic disease(s)
* Recent musculoskeletal injury handgrip exercise
* Prescription of chronic medications other than oral contraceptives
* History of hypertension or presence of arrhythmia

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Forearm blood flow | Baseline - Immediately before active and control interventions
  Doppler ultrasound - tested at rest and during rhythmic handgrip exercise with and without lower body negative pressure
Forearm blood flow | Immediately after active and control interventions (IPC only)
  Doppler ultrasound - tested at rest and during rhythmic handgrip exercise with and without lower body negative pressure
Forearm blood flow | 1 hour after active and control interventions (Diet intervention only)
  Doppler ultrasound - tested at rest and during rhythmic handgrip exercise with and without lower body negative pressure
Forearm blood flow | 2 hours after active and control interventions (Diet intervention only)
  Doppler ultrasound - tested at rest and during rhythmic handgrip exercise with and without lower body negative pressure
Forearm blood flow | 3 hours after active and control interventions (Diet intervention only)
  Doppler ultrasound - tested at rest and during rhythmic handgrip exercise with and without lower body negative pressure
Forearm vascular conductance | Baseline - Immediately before active and control interventions
  Blood flow divided by blood pressure - tested at rest and during rhythmic handgrip exercise with and without lower body negative pressure
Forearm vascular conductance | Immediately after active and control interventions (IPC only)
  Blood flow divided by blood pressure - tested at rest and during rhythmic handgrip exercise with and without lower body negative pressure
Forearm vascular conductance | 1 hour after active and control interventions (Diet intervention only)
  Blood flow divided by blood pressure - tested at rest and during rhythmic handgrip exercise with and without lower body negative pressure
Forearm vascular conductance | 2 hours after active and control interventions (Diet intervention only)
  Blood flow divided by blood pressure - tested at rest and during rhythmic handgrip exercise with and without lower body negative pressure
Forearm vascular conductance | 3 hours after active and control interventions (Diet intervention only)
  Blood flow divided by blood pressure - tested at rest and during rhythmic handgrip exercise with and without lower body negative pressure

SECONDARY OUTCOMES:
Blood pressure | Baseline - Immediately before active and control interventions
  Finger plethysmography - tested at rest and during rhythmic handgrip exercise with and without lower body negative pressure
Blood pressure | Immediately after active and control interventions (IPC only)
  Finger plethysmography - tested at rest and during rhythmic handgrip exercise with and without lower body negative pressure
Blood pressure | 1 hour after active and control interventions (Diet intervention only)
  Finger plethysmography - tested at rest and during rhythmic handgrip exercise with and without lower body negative pressure
Blood pressure | 2 hours after active and control interventions (Diet intervention only)
  Finger plethysmography - tested at rest and during rhythmic handgrip exercise with and without lower body negative pressure
Blood pressure | 3 hours after active and control interventions (Diet intervention only)
  Finger plethysmography - tested at rest and during rhythmic handgrip exercise with and without lower body negative pressure
Heart rate | Baseline - Immediately before active and control interventions
  ECG - tested at rest and during rhythmic handgrip exercise with and without lower body negative pressure
Heart rate | Immediately after active and control interventions (IPC only)
  ECG - tested at rest and during rhythmic handgrip exercise with and without lower body negative pressure
Heart rate | 1 hour after active and control interventions (Diet intervention only)
  ECG - tested at rest and during rhythmic handgrip exercise with and without lower body negative pressure
Heart rate | 2 hours after active and control interventions (Diet intervention only)
  ECG - tested at rest and during rhythmic handgrip exercise with and without lower body negative pressure
Heart rate | 3 hours after active and control interventions (Diet intervention only)
  ECG - tested at rest and during rhythmic handgrip exercise with and without lower body negative pressure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Guelph - Human Cardiovascular Physiology Laboratory, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teixeira AL, Gangat A, Bommarito JC, Burr JF, Millar PJ. Ischemic Preconditioning Acutely Improves Functional Sympatholysis during Handgrip Exercise in Healthy Males but not Females. Med Sci Sports Exerc. 2023 Jul 1;55(7):1250-1257. doi: 10.1249/MSS.0000000000003148. Epub 2023 Feb 24. PMID 36878187